CLINICAL TRIAL: NCT00235274
Title: Effects of RG1068 (Secretin) on Information Processing in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Shekhar, Anantha M.D., Ph.D. (Individual); Repligen Corporation (Industry)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0507-30; 4587049
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Secretin
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Subcutaneous Secretin

SUMMARY:
The overarching purpose of the proposed study is to determine Secretin's (RG1068) psychophysiological effects on measures of motor learning, affective, and inhibitory information processing in individuals with schizophrenia. Motor learning will be assessed with a classical eye-blink conditioning procedure, requiring the learning of a reflexive eye-blink response to a weak puff of air to the eye.

DETAILED DESCRIPTION:
In a recent placebo-controlled, double-blind, multicenter study of Secretin in refractory schizophrenics, we found that a patient who received Secretin (1.0 g/kg) intravenously, showed a marked improvement in eye blink conditioning following infusion. This subject also showed a clinical improvement of > 20% on the Total Score and Total Negative Score of the Positive and Negative Syndrome Scale (PANSS). Therefore, the primary objective of this study is to confirm and extend this observation in a larger group of individuals with schizophrenia. In this 24 to 48 hour experiment, the acquisition and extinction of the conditioned blink response will be assessed in participants with schizophrenia who are randomly assigned to one of two double blind treatment groups: (1) subcutaneous saline or (2) subcutaneous Secretin (20 ug/kg). Enrolled participants will remain on their stable medication regime (i.e., psychotropic medications and related treatments will not be manipulated). Furthermore, given evidence that Secretin administration increases the amygdala's activation during experimental presentation of fear-related facial cue stimuli, we wish to also investigate the effects of the experimental agent on psychophysiological processes putatively related to amygdala function. Prepulse inhibition is a widely studied paradigm in the schizophrenia literature, thought to reflect disruption of early sensory-motor gating that is present in both individuals with schizophrenia and their unaffected biological relatives, and can be mediated by various limbic structures including the amygdala. Therefore, as a secondary aim, the effects of Secretin will be tested on affect modulation, pre-pulse inhibition, and pre-pulse facilitation of the acoustic startle response using common psychophysiological research procedures. These procedures are frequently used in our laboratory and are currently approved for our use by the IRBs at both IUPUI and IUB.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent
2. DSM-IV diagnosis of schizophrenia
3. 18-55 years of age
4. Stable medication > 4 weeks

Exclusion Criteria:

1. Active suicidal ideation
2. Concurrent DSM-IV comorbidity with any substance dependence
3. A urine drug screen that is qualitatively positive for controlled substances
4. Abnormal hepatic function (AST or ALT > 2.5 X the upper limit of normal, or bilirubin > 1.5 X the upper limit of normal)
5. Abnormal renal function (BUN or creatinine > 1.5 X the upper limit of normal)
6. Abnormal bone marrow function (WBC < 4 x 103/mm3, Platelets <100 x 103/mm3 and hemoglobin <10 g/dl)
7. Any history of sensitivity to any of the ingredients in the study drug
8. Clinically significant organic disease including cardiovascular, hepatic, pulmonary, neurologic, or renal disease or other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the Investigator, would interfere with the performance or interpretability of, or put the patient at risk from, the study procedures.
9. Women who are pregnant, breastfeeding, or refuse to use adequate birth control

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-11; Study Completion 2006-08

PRIMARY OUTCOMES:
Motor learning will be assessed with a classical eye-blink conditioning procedure, requiring the learning of a reflexive eye-blink response to a weak puff of air to the eye.

SECONDARY OUTCOMES:
Effects of Secretin will be tested on affect modulation, pre-pulse inhibition, and pre-pulse facilitation of the acoustic startle response using common psychophysiological research procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Anantha Shekhar, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- LaRue Carter Hospital, Indianapolis, Indiana, United States